CLINICAL TRIAL: NCT03506776
Title: Foot Intervention Study Utilizing Commercially Available Infrared Thermometers With Individuals With Diabetes Using a Mixed Methods Approach
Brief Title: Foot Intervention Study Utilizing Commercially Available Infrared Thermometers With Individuals With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Collaborators: Health Care Foundation, NL, Canada (Unknown); Association of Registered Nurses of Newfoundland and Labrador (Unknown); NL-SUPPORT, NL, Canada (Unknown)
Responsible Party: Principal Investigator, Kathleen Stevens, Assistant Professor, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MemorialUN
Record Dates: First submitted 2018-03-28; First posted 2018-04-24 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Only Group (Active Comparator): The education only group will receive foot self-management education.
  Interventions: Other: Education Only Group
- Education and Thermometer Group (Experimental): The intervention group will receive foot self-management education. Additionally, the intervention group will receive a Commercially Available Infrared Thermometer (CAIT). Education on use of the CAIT will be provided through demonstration using a foot model and CAIT.
  Interventions: Device: Education and Thermometer Group

INTERVENTIONS:
Device: Education and Thermometer Group — The education will be provided in video format utilizing the Canadian Association of Wound Care (CAWC) diabetic foot management YouTube video and one-on-one teaching. Participants will be provided with an inspection mirror with an extendable handle to assist with visualizing the bottom of the feet and a pedometer to measure daily activity. One-on-one teaching with the thermometer will be provided. Participants will be given a handout for reference on using the thermometer. The foot model will be marked with a zigzag pattern on the plantar surface to illustrate the path that should be used when measuring temperature. The support person will be included in the teaching if he/she will be assisting the participant to obtain temperature readings.
  Other Names: Infrared Thermometer
  Arms: Education and Thermometer Group
Other: Education Only Group — The education will be provided in video format utilizing the Canadian Association of Wound Care (CAWC) diabetic foot management YouTube video and one-on-one teaching. Participants will be provided with an inspection mirror with an extendable handle to assist with visualizing the bottom of the feet and a pedometer to measure daily activity.
  Arms: Education Only Group

SUMMARY:
Foot self-management is important in preventing diabetic foot ulcers. However, even when individuals care for their feet, the signs of inflammation are often missed. A tool that will identify inflammation, a sign of initial tissue damage, may be needed. Previous research has shown that foot temperature self-monitoring reduced ulcer incidence by providing a warning sign of inflammation. However, these studies used an expensive medical thermometer. The objectives for this mixed-methods study are: (1) to determine if a foot health intervention that utilizes an inexpensive commercially-available infrared thermometer (CAIT) improves foot outcomes for individuals with diabetes; (2) to identify factors impacting foot self-management; (3) and to explore the participants', family and support persons', and healthcare providers' experiences with foot self-management and the intervention. This study will have three phases: Phase 1, patients, family and support person, and healthcare providers will share their insights regarding foot self-management to inform the intervention; Phase 2, a six-month RCT will assess the effectiveness of a CAIT; Phase 3, interviews will be conducted with participants, family and support persons, and health providers to explore their experiences with the intervention.

DETAILED DESCRIPTION:
Diabetes is a global health emergency, which is estimated to increase throughout the 21st century (Guariguata et al., 2014). The prevalence of diabetes in Canada is increasing; in 2014, 6.7% of Canadians and 9% of Newfoundlanders and Labradorians had diabetes (Statistics Canada, 2014). In 2020 the number of people in Canada with diabetes is expected to rise to 2.5 million people, or 9.9% of the population (Canadian Diabetes Association, 2009).

Patients with diabetes are at risk for poor foot health and the estimated lifetime incidence of a diabetic foot ulcer (DFU) for this population is 25% (Singh, Armstrong, & Lipsky, 2005). In Canada in 2011 DFUs and related care cost the healthcare system 547 million dollars (Hopkins, Burke, Harlock, Jegathisawaran, & Goeree, 2015). Complicated DFUs that do not heal can lead to amputation; an estimated 85% of amputations are the result of a DFU (Canadian Association of Wound Care, 2015).

The increasing number of people with diabetes will result in a rise in foot complications such as DFUs (Canadian Diabetes Association, 2009). Therefore, it is important to develop strategies for the prevention of DFUs. An important aspect of maintaining foot health is self-management (Boulton et al., 2008; Chang, Peng, Chang, & Chen, 2013). However, there is limited literature related to the experiences of diabetic patients with foot management (Delea et al., 2015). As a result, little is known of the factors that need to be addressed to ensure successful uptake of a self-management strategy. Further exploration of the issue of foot self-assessment and self-management with patients and health care providers is needed in order to develop and implement effective and sustainable interventions.

Interventions to prevent DFUs need to provide patients with strategies to prevent skin breakdown. Due to neuropathy individuals with diabetes do not recognize the inflammation that occurs prior to skin breakdown. In many instances, by the time individuals have identified a problem the ulceration had already occurred (Lavery et al., 2004). For patients with diabetes factors such as pressure can contribute to inflammation and increase plantar foot temperature. Commercially available-infrared thermometers (CAITs) can be used to detect this temperature increase before skin breakdown. Once the increase is identified, the individual can relieve pressure, for example by resting, until the temperature normalizes and inflammation decreases. If the temperature does not normalize in two days then a physician should be consulted. Therefore, self-management strategies that focus on identifying and addressing early signs of inflammation, such as a temperature increase, may be effective in preventing skin breakdown.

Various systematic reviews, which contained three randomized control trials (RCTs), have indicated that the use of personal temperature monitoring with a medical grade thermometer was an effective way to predict, and thus prevent DFUs (Arad, Fonseca, Peters, & Vinik, 2011; Houghton, Bower, & Chant, 2013; van Netten et al., 2015). These thermometers cost approximately $700, which can be prohibitively expensive. A recent study compared inexpensive CAITs, that cost under $100, to medical infrared thermometers and found them to be a reliable measure of skin temperature (Mufti, Coutts, & Sibbald, 2015). However, this technology has not been used as part of an intervention and it is unknown if the CAIT will result in the same positive results as the medical grade thermometer. This study will fill this empirical gap.

The Canadian Diabetes Association's position statement on amputation prevention calls for affordable and timely access to devices, education, and care (Canadian Diabetes Association., 2015). Use of a CAIT may potentially meet this need and offers a low-cost self-management tool to prevent skin breakdown. The purpose of this mixed-methods study is to determine if a self-management strategy that utilizes a low-cost CAIT is effective to prevent DFUs. Through engagement with patients and healthcare providers this research will also examine factors impacting self-management not addressed in prior studies and utilize this information to inform the intervention.

Phase 1 (Qualitative) Purposive convenience sampling will be utilized in Phase 1 and patients, support persons, and healthcare providers will be selected that will inform the researcher about issues with foot self-management. To gain a comprehensive understanding of foot self-management, participants will be selected who have a variety of experiences and characteristics, such as patients with diabetes with various foot health challenges and healthcare providers with different professional designations such as physicians and nurses. Semi-structured interviews lasting 20-30 minutes will be conducted at a mutually convenient location over six-weeks. All interviews will be recorded, transcribed verbatim, and analyzed using content analysis to identify themes and recommendations for the intervention. For example, a finding from Phase 1 may be that patients are not sure what information to communicate to their healthcare provider about their feet. Such a finding would be addressed by incorporating into the intervention further education about communication and potentially a checklist that the patients can use to take with them for appointments.

Phase 2 (RCT) Using a list of randomly generated numbers patients will be assigned to the intervention or control group. The control group and intervention group will receive foot self-management education. The content of the education will be finalized following completion of Phase 1. The education will be provided in video format utilizing the Canadian Association of Wound Care (CAWC) diabetic foot management YouTube video and one-on-one teaching. Both groups will be provided with an inspection mirror with an extendable handle to assist with visualizing the bottom of the feet and a pedometer to measure daily activity. Additionally, the intervention group will receive a CAIT. Education on use of the CAIT will be provided through demonstration using a foot model and CAIT. The foot model will be marked with a zigzag pattern on the plantar surface to illustrate the path that should be used when measuring temperature. The support person will be included in the teaching if he/she will be assisting the participant to obtain temperature readings. The participant will also be provided with a letter explaining the study to take to his/her healthcare provider.

Data collection is the same for both groups with the addition of foot temperature measurement for the intervention group. The initial one-hour intake session will take place in the participant's home or at Memorial University School of Nursing and will include completing baseline assessments and distributing requisitions for bloodwork and the orthotic assessment, log books, and equipment. Use of one trained interviewer will minimize information bias during data collection.

At the end of the initial visit a second 15-minute visit will be booked with participants in the intervention group for one week later. The purpose of the second visit will be to determine if the thermometer is being used correctly and the documentation is being completed as intended. This will also be an opportunity to answer any questions. Next, the RA or researcher will contact the participant and support persons one week later (e.g.,, week 2) via phone to check if there are any questions or concerns. If the participant's concerns cannot be answered over the phone the RA or investigator will book a time to visit the participant. The log books for participants in the control group and intervention group will be picked up on a monthly basis either by the investigator or RA. A tracking form will be used to organize the timeframe for the phone calls and visits. Participants in the control group will be contacted via phone one week after the initial visit to address any questions or concerns. At three months and six months another hour-long appointment will be made with all participants to complete assessments and questionnaires.

If a participant develops an ulcer during the RCT his/her participation in the study will end but data collected will be included. A participant will be advised to immediately contact his/her physician if an area of concern is identified. Also, a participant will be asked to contact the investigator if he/she develops an ulcer.

The primary outcome is incidence of ulceration measured through physical assessment and self-report utilizing a standard definition of DFU. Secondary outcomes include any other foot-related changes, changes in satisfaction, quality of life, and self-efficacy. Confounding variables include: pedometer readings, HbA1C, orthotic assessment, temperature, depression symptoms, foot care behaviors, and information collected in the participant profile.

Phase 3 (Qualitative) At the end of the data collection of Phase 2 participants will be recruited for Phase 3. Semi-structured interviews will be conducted with 25 RCT participants (15 participants from the intervention group, 5 participants and their support person who assisted with measuring the foot temperature, 5 participants from the control group) and 10 healthcare providers who were consulted by participants during the intervention to obtain information about the experiences with self-management and the intervention. The interview with the participants and healthcare providers will be of 30-45 minutes duration and will take place at a mutually convenient location. The interviews with the support person will be conducted separately from the participant and will be of 20 minutes in duration. All interviews will be recorded and transcribed verbatim. The details of the methods, including the analysis that will be utilized in phase 3, will be developed after the completion of phase 2.

ELIGIBILITY:
Healthcare Providers (Phase 1 and 3)

Inclusion criteria are:

1. Provide care to diabetic individuals (Phase 1 only)
2. Work in one of the following areas: Eastern Health Diabetes Centre, Wound Care Clinic, and Community Health St. John's Region; Family Physician Clinics; Nurse Practitioner Clinics; and Podiatry Clinics (Phase 1 only)
3. Were consulted by participants during the intervention (Phase 3 only)

Patients (All Phases)

Inclusion criteria are:

1. Able to read and speak English
2. Reachable by telephone
3. 18 years of age and older
4. History fits with International Diabetic Foot Risk Classification System category 2 (decreased sensation and blood supply or foot deformity) or category 3 (previous ulcer or amputation) (Peters, 2005).

Inclusion criteria (Phase 2)

1. Callus and/or
2. Deformity and/or
3. One areas of loss of sensation as determined by assessment with Semmes Weinstein Monofilament

Exclusion criteria are:

1. Ulcer
2. Amputation sites not healed
3. Foot infections
4. Charcot arthropathy
5. Pregnancy and/or breastfeeding (pregnancy causes changes to feet; these women may find the demands of the study too great in consideration of the life changes they are experiencing)
6. Major health conditions
7. Inability to read the thermometer and no support person available to assist the participant with temperature reading and documentation on a daily basis
8. Severe peripheral vascular disease (PVD), as evidenced by non-palpable pulses or an ankle brachial index of < 0.7 on either extremity (Armstrong et al., 2007)
9. Unable to walk without assistance.

Family/Support Persons (Phase 1 and 3)

Inclusion criteria are:

1. 18 years of age and older (Phase 1 and 3).
2. Able to read and speak English (Phase 1 and 3).
3. Reachable by telephone (Phase 1 and 3).
4. Provides frequent tangible support to an individual with diabetes such as assisting with activities of daily living (Phase 1 and 3).
5. Assisted a participant during Phase 2 of the study (Phase 3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
change from baseline foot assessment as evidenced by a diabetic foot ulcer | time to ulceration up to 24 weeks
  Screening for the high risk diabetic foot: A 60 second foot tool (2012) Sibbald

SECONDARY OUTCOMES:
change from baseline foot assessment as evidenced by presence or absence of skin breakdown | Completed by participant daily up to 24 weeks
  Foot Assessment Log completed by participant
change from baseline foot assessment evidenced by presence or absence of redness | Completed by participant daily up to 24 weeks
  Foot Assessment Log completed by participant

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Stevens, PhD(c), Principal Investigator — Memorial University of Newfoundland and Labrador
Locations (1):
- Memorial University, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guariguata L, Whiting DR, Hambleton I, Beagley J, Linnenkamp U, Shaw JE. Global estimates of diabetes prevalence for 2013 and projections for 2035. Diabetes Res Clin Pract. 2014 Feb;103(2):137-49. doi: 10.1016/j.diabres.2013.11.002. Epub 2013 Dec 1. PMID 24630390
- [Background] Statistics Canada. Diabetes by age group and sex [table]. http://Www.statcan.gc.ca/tables-tableaux/sum-som/l01/cst01/health53a-eng.htm. 2014.
- [Background] Canadian Diabetes Association. Economic tsunami: The cost of diabetes in canada. www.diabetes.ca/publications-newsletters/advocacy-reports/economic-tsunami-the-cost-of-diabetes-in-canada; . 2009.
- [Background] Singh N, Armstrong DG, Lipsky BA. Preventing foot ulcers in patients with diabetes. JAMA. 2005 Jan 12;293(2):217-28. doi: 10.1001/jama.293.2.217. PMID 15644549
- [Background] Hopkins RB, Burke N, Harlock J, Jegathisawaran J, Goeree R. Economic burden of illness associated with diabetic foot ulcers in Canada. BMC Health Serv Res. 2015 Jan 22;15:13. doi: 10.1186/s12913-015-0687-5. PMID 25608648
- [Background] Canadian Association of Wound Care. Statistics. http://Cawc.net/index.php/public/facts-stats-and-tools/statistics/. 2015.
- [Background] Boulton AJ, Armstrong DG, Albert SF, Frykberg RG, Hellman R, Kirkman MS, Lavery LA, Lemaster JW, Mills JL Sr, Mueller MJ, Sheehan P, Wukich DK; American Diabetes Association; American Association of Clinical Endocrinologists. Comprehensive foot examination and risk assessment: a report of the task force of the foot care interest group of the American Diabetes Association, with endorsement by the American Association of Clinical Endocrinologists. Diabetes Care. 2008 Aug;31(8):1679-85. doi: 10.2337/dc08-9021. No abstract available. PMID 18663232
- [Background] Chang CH, Peng YS, Chang CC, Chen MY. Useful screening tools for preventing foot problems of diabetics in rural areas: a cross-sectional study. BMC Public Health. 2013 Jun 27;13:612. doi: 10.1186/1471-2458-13-612. PMID 23802741
- [Background] Delea S, Buckley C, Hanrahan A, McGreal G, Desmond D, McHugh S. Management of diabetic foot disease and amputation in the Irish health system: a qualitative study of patients' attitudes and experiences with health services. BMC Health Serv Res. 2015 Jul 1;15:251. doi: 10.1186/s12913-015-0926-9. PMID 26129712
- [Background] Lavery LA, Higgins KR, Lanctot DR, Constantinides GP, Zamorano RG, Armstrong DG, Athanasiou KA, Agrawal CM. Home monitoring of foot skin temperatures to prevent ulceration. Diabetes Care. 2004 Nov;27(11):2642-7. doi: 10.2337/diacare.27.11.2642. PMID 15504999
- [Background] Arad Y, Fonseca V, Peters A, Vinik A. Beyond the monofilament for the insensate diabetic foot: a systematic review of randomized trials to prevent the occurrence of plantar foot ulcers in patients with diabetes. Diabetes Care. 2011 Apr;34(4):1041-6. doi: 10.2337/dc10-1666. No abstract available. PMID 21447666
- [Background] Houghton VJ, Bower VM, Chant DC. Is an increase in skin temperature predictive of neuropathic foot ulceration in people with diabetes? A systematic review and meta-analysis. J Foot Ankle Res. 2013 Aug 7;6(1):31. doi: 10.1186/1757-1146-6-31. PMID 23919736
- [Background] van Netten JJ, Price PE, Lavery LA, Monteiro-Soares M, Rasmussen A, Jubiz Y, Bus SA; International Working Group on the Diabetic Foot. Prevention of foot ulcers in the at-risk patient with diabetes: a systematic review. Diabetes Metab Res Rev. 2016 Jan;32 Suppl 1:84-98. doi: 10.1002/dmrr.2701. PMID 26340966
- [Background] Mufti A, Coutts P, Sibbald RG. Validation of commercially available infrared thermometers for measuring skin surface temperature associated with deep and surrounding wound infection. Adv Skin Wound Care. 2015 Jan;28(1):11-6. doi: 10.1097/01.ASW.0000459039.81701.b2. PMID 25502971
- [Background] Canadian Diabetes Association. Canadian diabetes association's position statement on amputation prevention.http://Www.diabetes.ca/about-cda/public-policy-position-statements/amputation-prevention. 2015.
- [Background] Lavery LA, Higgins KR, Lanctot DR, Constantinides GP, Zamorano RG, Athanasiou KA, Armstrong DG, Agrawal CM. Preventing diabetic foot ulcer recurrence in high-risk patients: use of temperature monitoring as a self-assessment tool. Diabetes Care. 2007 Jan;30(1):14-20. doi: 10.2337/dc06-1600. PMID 17192326
- [Background] Armstrong DG, Holtz-Neiderer K, Wendel C, Mohler MJ, Kimbriel HR, Lavery LA. Skin temperature monitoring reduces the risk for diabetic foot ulceration in high-risk patients. Am J Med. 2007 Dec;120(12):1042-6. doi: 10.1016/j.amjmed.2007.06.028. PMID 18060924